CLINICAL TRIAL: NCT04147130
Title: Efectiveness of the MultiPAP Plus Intervention in Young-old Patients With Multimorbidity and Polypharmacy Aimed at Improving Prescription in Primary Care: Cluster RCT
Brief Title: MultiPAP Plus: Improving Prescription in Primary Care Patients With Multimorbidity and Polypharmacy
Acronym: MultiPAP Plus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Aragones de Ciencias de la Salud (Other Government)
Collaborators: Gerencia de Atención Primaria, Madrid (Other Government); Aragon Institute for Health Research (IIS Aragón) (Unknown); Andaluz Health Service (Other Government); Fundación de Investigación e Innovación Biomédica Atención Primaria (FIIBAP) (Unknown); Red de Investigación en Servicios de Salud en Enfermedades Crónicas (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Principal Investigator, Alexandra Prados Torres, Principal Investigator, MD, PhD, Instituto Aragones de Ciencias de la Salud
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: PI 18/01303,18/01515,18/01812
Record Dates: First submitted 2019-10-22; First posted 2019-10-31 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Multimorbidity; Polypharmacy; Comorbidities and Coexisting Conditions; Clinical Decision-Support Systems
Keywords: Primary Health Care; Medication Adherence; Disability; Patient-Centered Care; Ariadne Principles
MeSH Terms: conditions — Medication Adherence

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MultiPAP Plus intervention (Experimental): Complex intervention with general practitioners and patients
  Interventions: Other: MultiPAP Plus; Other: Usual care
- Usual care (Active Comparator): Patients will recieve the usual clinical care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: MultiPAP Plus — Complex intervention incorporating previous MultiPAP intervention (based on the ARIADNE principles with two main components: 1) Training of general practitioners and 2) Patient-centered clinical interview) And it adds a clinical-decision support system to help structured treatment-plan review.
  Arms: MultiPAP Plus intervention
Other: Usual care — Patients will receive the usual clinical care based on current clinical practice guidelines.

SUMMARY:
This study assesses the effectiveness of a complex intervention in young-old patients with multimorbidity and polypharmacy aimed at improving physician drug prescription in primary care, measured by hospitalization-mortality at six 6 (T1), 12 (T2) and 18 (T3) months from baseline compared to usual care.

DETAILED DESCRIPTION:
Design: Pragmatic cluster randomized clinical trial with 18 months follow-up.

Unit of randomization: general practitioner.

Unit of analysis: patient.

Setting: Primary Health Care Centres in three different Spanish Autonomous Communities (Aragón, Madrid and Andalucía).

Population: Patients 65-74 years of age with multimorbidity (3 or more chronic diseases) and polypharmacy (5 or more drugs taken for at least three months). N=1234 patients (617 in each arm, 8 patients per physician) will be recruited by general practitioners before randomization.

Intervention: Complex intervention incorporating previous MultiPAP intervention (based on the ARIADNE principles with two main components: 1) Training of general practitioners and 2) Patient-centered clinical interview) And it adds a clinical-decision support system to help structured treatment-plan review.

Control group: usual care.

Variables: First level (Patient): a) Main: hospitalizations and/or mortality; b) Secondary: health services use, quality of life (Euroqol 5D-5L), disability (WHODAS), fractures, pharmacotherapy and adherence to treatment (Morisky-Green), clinical and socio-demographic. Second level (Physician): a) Socio-demographic. b) CDSS use: acceptance and satisfaction of health care provider use c) Professional background: time in the position, center characteristics and medical education involvement.

Analysis: All analyses will be carried out adhering to the intention-to-treat principle. Description of baseline characteristics. Basal comparison between groups. Analysis of primary outcome: difference in percentages in the final combined variable from 0 (T0) to 18 months (T3), with its corresponding 95% CI. Adjustement by main confounding and prognostic factors will be performed through a multilevel analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients 65-74 years of age with multimorbidity (3 or more chronic diseases) and polypharmacy (5 or more drugs taken for at least three months).
* Informed consent.

Exclusion Criteria:

* Institutionalized patient at nursing homes or similar
* Life expectancy < 12 months

Ages: 65 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1162 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Hospitalizations and/or mortality | From Baseline to Month 18
  Difference in percentages in the final combined variable

SECONDARY OUTCOMES:
Hospitalizations and/or mortality (T2) | From Baseline to Month 12
  Difference in percentages in the final combined variable
Therapeutic adherence questionnaire | Baseline, 6, 12 and 18 months
  Morisky-Green questionnaire. Dicotomous variable. Any wrong answer to any of the four questions would mean worse adherence
Medication Safety: Potentially Drug-Drug interactions (DDI), Potentially Innappropiate Medication (PIM), Adverse Drug Reactions | Baseline, 6, 12 and 18 months
  Number of Potentially Drug-Drug interactions (DDI) per patient, Number of Potentially Innappropiate Medication (PIM) per patient, Number of Adverse Drug Reactions per patient
Use of health services | at 12 and at 18 months
  Number of Unscheduled and/or avoidable hospitalizations, number of visits to emergency services and primary care (Family Physician and nurse).
Disability | Baseline, 12 and 18 months
  World Health Organization Disabilty Assessment (WHODAS). 12-items abbreviated scale (0=No Difficulty, 1=Mild Difficulty, 2=Moderate Difficulty, 3=Severe Difficulty, and 4=Extreme Difficulty or Cannot Do). Maximum 48 points.
Perceived Quality of Life: Euroqol 5D-5L questionnaire | Baseline, 12 and 18 months
  EQ5D is one of the most widely used health states descriptive system and has a valuation in Spain.
  EQ-5D questionnaires have 5 dimensions: "Mobility", "Human Autonomy," "Current Activities", "Pain / Discomfort", "Anxiety / Depression" and all dimensions are described by 5 problem levels corresponding to patient response choices.
  A quality of life score is obtained according to the answers to the questionnaires.
System Usability Scale of the CDSS | at 6 and 18 months.
  It consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Alexandra Prados-Torres, MD,PhD, Principal Investigator — Instituto Aragonés de Ciencias de la Salud (IACS); Daniel Prados-Torres, MD, PhD, Principal Investigator — Servicio Andaluz de Salud (Andaluz Health Service); Isabel Del Cura-González, MD,PhD, Principal Investigator — Gerencia Asistencial de Atención Primaria, Madrid
Locations (3):
- Spain (3):
  - Servicio Andaluz de Salud, Málaga, Andalusia
  - Instituto Aragonés de Ciencias de la Salud (IACS), Zaragoza, Aragon
  - Gerencia Asistencial de Atención Primaria de Madrid, Madrid

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Del Cura-Gonzalez I, Lopez-Rodriguez JA, Leiva-Fernandez F, Gimeno-Feliu LA, Pico-Soler V, Bujalance-Zafra MJ, Dominguez-Santaella M, Polentinos-Castro E, Poblador-Plou B, Ara-Bardaji P, Aza-Pascual-Salcedo M, Rogero-Blanco M, Castillo-Jimenez M, Lozano-Hernandez C, Gimeno-Miguel A, Gonzalez-Rubio F, Medina-Garcia R, Gonzalez-Hevilla A, Gil-Conesa M, Martin-Fernandez J, Valderas JM, Marengoni A, Muth C, Prados-Torres JD, Prados-Torres A; MULTIPAP PLUS Group. Effectiveness of the MULTIPAP Plus intervention in youngest-old patients with multimorbidity and polypharmacy aimed at improving prescribing practices in primary care: study protocol of a cluster randomized trial. Trials. 2022 Jun 9;23(1):479. doi: 10.1186/s13063-022-06293-x. PMID 35681224